CLINICAL TRIAL: NCT06518694
Title: Beta-blOckers discoNtinuation in Patients Presenting Heart FaIlure With REcovered Left Ventricular Ejection Fraction
Acronym: BONFIRE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: APHP230833; P-PHRC-22-0112 (Other Grant/Funding Number: Direction générale de l'offre de soins[DGOS])
Record Dates: First submitted 2024-06-21; First posted 2024-07-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart Failure relapse; Recovered Ejection Fraction; Cardiovascular outcomes; Hospitalization for CV reason; Death; Bisoprolol; Carvedilol; Metoprolol; Nebivolol; Randomized
MeSH Terms: conditions — Heart Failure; Death

STUDY DESIGN:
Intervention Model Description: National, Multicenter, Randomised, Open-label, Non-inferiority, Blinded endpoints prospective trial
Who Masked: Outcomes Assessor
Masking Description: Only outcomes assessor will be blinded to the study arm (Blinded endpoints prospective trial)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): Βeta-Blockers therapy will be discontinued (with tapering) while the remaining guideline-directed optimal medical therapy for HF is maintained
  Interventions: Drug: Βeta-Blockers discontinued (with tapering)
- Group2 (No Intervention): The patients will continue their usual guideline-directed optimal medical therapy for HF, including Βeta-Blockers therapy, without modification.

INTERVENTIONS:
Drug: Βeta-Blockers discontinued (with tapering) — The experimental group will undergo discontinuation of their beta-blockers treatment during the study period.
  The tapering of beta-blocker will start on the day after randomisation and is based on a reduction by half-dose every 48 hours (1/2 maximally recommended dose for 48 hours, then ¼ maximally recommended dose for 48 hours) until reaching the minimal recommended dosage (1/8 maximally recommended dose) for 48 hours before complete interruption of treatment. Consequently, the tapering will not be needed in patients already receiving the minimal recommended dosage (i.e., 1/8 dose) at inclusion, and these patients will be instructed to stop taking beta-blockers the day after randomisation.
  Arms: Group1

SUMMARY:
A significant proportion of patients initially diagnosed with heart failure and a reduced left ventricular ejection fraction (LVEF<40%, HFrEF) presents a substantial improvement in response to evidence-based medical and device therapies. Some of these patients (estimated from 20 to 30%) even display a complete normalization of LVEF (i.e., >50%) and are now recognized as a specific sub-group of patients named Heart Failure with recovered Ejection Fraction (HFrecovEF). Different studies have shown that reverse remodeling with recovery of cardiac function and stabilization of HF symptoms are associated with improved clinical outcomes over the long-term. Whether these patients present a stable remission of HF and could benefit a therapeutic de-escalation is however unclear. Until novel data are provided, medical therapies are thus continued indefinitely in these stable patients with HFrecovEF. Current guidelines for the management of patients with heart failure and a reduced left ventricular ejection fraction recommends a comprehensive therapy, including 5 different therapeutic classes (RAAS blockers (with a preference for ARNi) + Beta-Blockers + SGLT2i + Mineraloreceptors Antagonists + or - Diuretics ).

None of these therapies (with the recent exception of one SGLT2i, i.e. Dapagliflozin) have been tested in patients with HFrecovEF. In addition, it is unclear whether the benefit of older therapies (notably beta-blockers) remains in patients receiving modern comprehensive therapy as newer drugs were tested as add-on therapies. This polypharmacy is lowering adherence and is creating a challenge for physicians and patients. Betablockers are notably associated with frequent side effects, a limited tolerance and a significant reduction of quality of life. Their efficacy on outcomes is not established in patients with normal LVEF. Pilot studies have suggested that Beta-blockers interruption in patients with HF and normal EF was associated with functional improvement.

DETAILED DESCRIPTION:
BONFIRE is a National, Multicenter, Randomised, Open-label, Non-inferiority, Blinded endpoints prospective trial.

The study concerns HF patients with a history of reduced left ventricular ejection fraction (45% or below), but with a normalized LVEF (currently ≥ 50 % on cardiac echography) under an optimal medical therapy as recommended in European guidelines (including beta-blockers, RAAS blockade with ARNI or ACE-I or ARBs, SGLT2 inhibitors, MRA, + or - loop diuretics) AND with no or mild symptoms and no heart failure-related events within the last six months.

The patients fulfilling the full inclusion criteria and without exclusion criteria, that agree to participate the protocol and that have signed the informed consent will be randomized (1:1) into two groups:

* Experimental group (N=650): Βeta-Blockers therapy will be discontinued (with tapering) while the remaining guideline-directed optimal medical therapy for HF is maintained.
* Control group (N=650): The patients will continue their usual guideline-directed optimal medical therapy for HF, including Βeta-Blockers therapy, without modification.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years-old
2. Established diagnosis of HF for more than 12 months, from an ischemic or a non-ischemic origin
3. With a documented history of reduced left ventricular ejection fraction (LVEF ≤ 45%), followed by a normalisation of LVEF (≥ 50 % for the last 6 months) assessed by cardiac echography.
4. With a left ventricular end diastolic volume indexed to body surface area (LVEDVi) within the normal range (≤74ml/m2 in men and ≤61 ml/m2 in women)
5. No or mild symptoms of HF (defined as NYHA functional class I or II)
6. No heart failure-related hospital admission within the last six months
7. Currently receiving a beta-blocker indicated for chronic heart failure (i.e. bisoprolol or carvedilol or metoprolol or nebivolol) whatever the dose used, for at least 12 months
8. And receiving the guideline-directed optimal medical therapy for at least 12 months (i.e., maximal tolerated dose of SGLT2 inhibitors, and of RAAS blocker (Angiotensin receptor neprilysin inhibitor OR Angiotensin-converting-enzyme-inhibitors OR Angiotensin II receptors blockers), and MRA if tolerated). Loop diuretics use is adjusted to congestive signs according to physicians' decision.

   No initiation or major adjustment in heart failure therapies should have occurred during the 3 months prior to study inclusion.
9. With or without ICD
10. Ability to provide written informed consent to participate to the study
11. Patient affiliated to Social Security

Exclusion Criteria:

1. Atrial, supra-ventricular, or ventricular arrhythmias, in the last 12 months and/or requiring beta-blockers according to investigator.
2. Uncontrolled arterial hypertension according to investigator decision.
3. Symptomatic angina or evidence of infra-clinic myocardial ischemia requiring beta-blockers according to investigator decision.
4. Cardiac resynchronization therapy
5. Extra-cardiac conditions requiring beta-blockers (migraine, essential tremor, prevention of bleeding from esophageal varices in patients with liver cirrhosis, adrenergic symptoms of hyperthyroidism…) according to investigator decision.
6. History of severe outcomes at beta-blockers interruption: HF relapse, occurrence of arrythmias
7. Severe valvulopathy, restrictive, infiltrative or hypertrophic cardiomyopathy, constrictive pericarditis, or acute myocarditis within 3 months prior to inclusion Visit.
8. Planned coronary, carotid, or peripheral artery revascularization known at the day of inclusion
9. Chronic renal failure with eGFR <20mL/Min per 1.73m² (CKD-Epi) at inclusion
10. Hepatic insufficiency classified as Child-Pugh B or C at the inclusion Visit.
11. Any past solid organ transplantation or planned organ transplantation within 12 months
12. Any condition other than HF that could limit survival to less than one year
13. Pregnancy or breastfeeding women or women of childbearing potential without adequate contraceptive method
14. Current participation in another interventional trial.
15. Patient under legal protection (protection of the court, or in curatorship or guardianship).
16. Any disorder, unwillingness or inability, which in investigator's opinion, might jeopardise the patient's safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study will be evaluated with one-year minimum follow-up and will be the composite of: | Within 1 year minimum after randomization
  - HF relapse (at any time during the study period):
  * drop in LVEF >10% (expressed as absolute value)
  * relative increase in body surface area-indexed left ventricular end-diastolic volume (LVEDVi) >10%
  * increase in NT-proBNP >2x and ≥ 400 ng/L
  * worsening heart failure symptoms requiring hospitalization or urgent visits or out-of-hospital therapeutic management with diuretics (intra-venous or oral).
death | Within 1 year minimum after randomization
  All-cause death
Hospitalisation for CV reason | Within 1 year minimum after randomization
  - Hospitalisation for CV reason (ACS or need for coronary catheterization +/- revascularization / supra-ventricular arrhythmias / ventricular arrhythmias / Syncope, Pace-Maker implantation / High blood pressure / Stroke).

SECONDARY OUTCOMES:
HF relapse defined by: | At each visit from randomization through study completion, an average of 4 years
  * Reduction in LVEF by more than 10% (absolute value)
  * A relative increase in LVEDVi by more than 10%
  * A two-fold rise in baseline NT-pro-BNP concentration and to more than 400 ng/L.
  * Clinical evidence of heart failure, based on signs and symptoms as adjudicated by the research team.
  * Hospitalization for worsening HF
Death | At each visit from randomization through study completion, an average of 4 years
  All-cause Death
All individual reasons for Hospitalisation, as follows: | At each visit from randomization through study completion, an average of 4 years
  * ACS or need for coronary catheterisation +/-revascularization
  * Recurrent ischemia
  * Supra-ventricular or ventricular arrhythmias
  * Syncope, PM implantation
  * High blood pressure
  * Stroke
Cardiovascular death | At each visit from randomization through study completion, an average of 4 years
  All-cause cardiovascular death
Number of patients with reduction in LVEF | At each visit from randomization through study completion, an average of 4 years
  Number of patients with reduction in LVEF by more than 10% (absolute value) and to less than 50%.
Number of patients with a relative increase in LVEDVi | At each visit from randomization through study completion, an average of 4 years
  Number of patients with a relative increase in LVEDVi by more than 10% and to higher than the normal range.
Number of patients hospitalized | At each visit from randomization through study completion, an average of 4 years
  Number of patients hospitalized for worsening HF
Number of patients needing loop diuretics | At each visit from randomization through study completion, an average of 4 years
  Number of patients needing loop diuretics for congestive symptoms, during hospitalization and/or in out-of-hospital settings
Changes in NYHA Class | At each visit from randomization through study completion, an average of 4 years
  Changes in NYHA Class
Absolute values of NT-pro-BNP concentrations at the different visits | At each visit from randomization through study completion, an average of 4 years
  Absolute values of NT-pro-BNP concentrations at the different visits
Proportion of patients with changes in NT-proBNP concentrations to more than 400 ng/L. | At each visit from randomization through study completion, an average of 4 years
  Proportion of patients with changes in NT-proBNP concentrations to more than 400 ng/L.
Number of patients needing beta-blocker re-introduction in the experimental group or beta-blocker discontinuation in the control group | At each visit from randomization through study completion, an average of 4 years
  Number of patients needing beta-blocker re-introduction in the experimental group or beta-blocker discontinuation in the control group
Occurrence of arrhythmic events (any types, i.e., supra-ventricular and/or ventricular arrhythmias & requiring hospitalization or not) in all participants | At each visit from randomization through study completion, an average of 4 years
  Occurrence of arrhythmic events (any types, i.e., supra-ventricular and/or ventricular arrhythmias & requiring hospitalization or not) in all participants
Occurrence of infra-clinic supra-ventricular and/or ventricular arrhythmias in patients implanted with ICD before participating the study | At each visit from randomization through study completion, an average of 4 years
  Occurrence of infra-clinic supra-ventricular and/or ventricular arrhythmias in patients implanted with ICD before participating the study
Quality of life (QoL) evaluated by the auto-questionnaire (EQ5D) | At each visit from randomization through study completion, an average of 4 years
  Quality of life (QoL) evaluated by the auto-questionnaire (EQ5D)
Quality of life with heart failure, evaluated by the auto-questionnaire KCCQ-12 filled by the patients himself. | At each visit from randomization through study completion, an average of 4 years
  Quality of life with heart failure, evaluated by the auto-questionnaire KCCQ-12 filled by the patients himself.
Anxiety | At each visit from randomization through study completion, an average of 4 years
  questionnaire HADS (Hospital Anxiety and Depression Scale), score de 0 à 21, higher scores indicate the presence of anxiety or depression
Erectile dysfunction (in men only) | At each visit from randomization through study completion, an average of 4 years
  Erectile dysfunction (in men only) by the questionnaire IIEF5 (International Index of Erectile Function).
Absolute values of heart rate at the different visits | At each visit from randomization through study completion, an average of 4 years
  Absolute values of heart rate at the different visits and relative change as compared to baseline values (first year)
Evaluation of Side effects: Questionnaire on the Presence of Blury Vision | At each visit from randomization through study completion, an average of 4 years
  Questionnaire on the Presence of Blury Vision
Evaluation of Side effects: Sensation of cold hands and feet | At each visit from randomization through study completion, an average of 4 years
  Sensation of cold hands and feet
Evaluation of Side effects : Insomnia | At each visit from randomization through study completion, an average of 4 years
  Insomnia
Occurrence of Palpitations | At each visit from randomization through study completion, an average of 4 years
  Occurrence of Palpitations
Syncope / Dizziness requiring a consultation | At each visit from randomization through study completion, an average of 4 years
  Syncope / Dizziness requiring a consultation
Evaluation of adherence to therapies evaluated by self-questionnaire | At each visit from randomization through study completion, an average of 4 years
  Evaluation of adherence to therapies evaluated by self-questionnaire
Exercise capacity by 6M walk test (in participating centers) | At each visit from randomization through study completion, an average of 4 years
  Exercise capacity by 6M walk test (in participating centers)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Sébastien HULOT, MD,PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No